CLINICAL TRIAL: NCT06408792
Title: Randomized Controlled Tiral to Evaluate Postoperative Pain and Quality of Life in Relation to Oral Health After Taking a Deephethelized Gingival Graft and Covering it With an Adhesive Film of Cellulose and Fluid Composite in Comparison With a Palate Plate or Cyanocrylate.
Brief Title: To Evaluate Postoperative Pain and Quality of Life After Taking a Deephethelized Gingival Graft and Covering it With Different Treatments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24/175-EC_X
Record Dates: First submitted 2024-03-13; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Quality of Life; Palate; Wound
MeSH Terms: conditions — Pain, Postoperative; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cellulose (OraAid) and fluid composite (Experimental): In this case, collagen sponges will be placed in the palatal wound, then the cellulose adhesive film (OraAid) will be placed on top, and this will be covered by fluid composite adhered to the teeth on their palatal wall.
  Amoxicillin 750mg 1pill each 8hours during 7 days. Ibuprofen 600mg 1pill each 8hours when needed.
  Interventions: Device: Deepithelized graft and protection technique
- Palate plate (Active Comparator): In this case, collagen sponges will be placed in the palatal wound, held in place by sutures, and the palatal wound will be covered with a custom-made palatal plate made just after surgery.
  Amoxicillin 750mg 1pill each 8hours during 7 days. Ibuprofen 600mg 1pill each 8hours when needed.
  Interventions: Device: Deepithelized graft and protection technique
- Cyanocrylate (periacril) (Active Comparator): In this case, collagen sponges will be placed in the palatal wound held by sutures and the palatal wound will be covered with cyanoacrylate tissue adhesive (Periacryl 90).
  Amoxicillin 750mg 1pill each 8hours during 7 days. Ibuprofen 600mg 1pill each 8hours when needed.
  Interventions: Device: Deepithelized graft and protection technique

INTERVENTIONS:
Device: Deepithelized graft and protection technique — To obtain the graft in all cases, on the day of surgery, 4% articaine with epinephrine 1:100,000 will be administered to block the greater palatine nerve. Gingival grafts from all groups will be deepithelialized intraorally using a sterile 834 turbine diamond bur. This drill will go deeper into the palatal mucosa 0.5mm (half of the outermost active part of the drill). The gingival grafts will be obtained with the surgical technique described by Zucchelli et al. 2010.

SUMMARY:
Objective: To evaluate postoperative pain and quality of life in relation to oral health after obtaining a palatal de-epithelialized gingival graft and subsequent coverage of the surgical wound with an adhesive film of cellulose and fluid composite versus a palatal plate or covering with cyanoacrylate.

Study design: Randomized controlled study.

Patients: Patients who require a de-epithelialized gingival graft will be selected from two private clinics in the Community of Madrid.

Allocation: Patients will be randomly assigned to the study group (cellulose film and flowable composite), control group 1 (palatal plank) or control group 2 (cyanoacrylate coverage).

Variables: Postoperative pain will be recorded using a 10 cm visual analogue scale (VAS) and analgesic consumption will be noted. Quality of life in relation to oral health will be recorded using the Oral Health Impact Profile-14 (OHIP-14) questionnaire.

Analysis plan: Descriptive statistics will be used to describe patient characteristics. The possible differences between the 3 study groups will be evaluated using parametric or non-parametric tests depending on the distribution of the variables.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years.
2. Need for soft tissue augmentation in an edentulous space to increase gingival volume simultaneously with placing a dental implant.
3. Patients with a palatal thickness of at least 4mm. This will be measured by overlaying a DICOM file of the CBCT with an STL file of the intraoral scan (Shining 3D). It will be measured at the height of the maxillary 2nd premolar, 5mm from the gingival margin.
4. Patients in whom a de-epithelialized palatal graft measuring 12x5mm can be obtained and which is between 1.5-2mm thick. The thickness will be measured with a digital caliper once it has been de-epithelialized.
5. Patients with no history of previous palatal graft extraction.
6. Patients with the ability to comply with the procedures related to the study, such as maintaining good oral hygiene, filling out the questionnaires and attending follow-up appointments.
7. Patients with the ability to fully understand the nature of the proposed surgery and the ability to understand and sign the informed consent form.

Exclusion Criteria:

1. Presence of vertical bone dehiscence of >3mm in the buccal area of the edentulous space where the implant will be placed (assessed at the time of surgery).
2. Smokers of more than 10 cigarettes/day
3. Presence of untreated periodontitis.
4. Diabetics
5. Patients being treated with oral anticoagulants or antiplatelet agents.
6. Patients with a history of malignant tumors, head and neck radiotherapy, chemotherapy or immunotherapy treatment in the last 5 years.
7. Patients with a history of previous or current medication that affects wound healing or promotes the appearance of infections, such as the use of corticosteroids, immunosuppressants or immunomodulators.
8. Patients with diseases that affect the metabolism of connective tissue, autoimmune or chronic inflammatory diseases with oral involvement (oral lichen planus, mucosal pemphigoid, pemphigus...), alterations in vascularization in the donor or recipient area, metabolic bone diseases or abuse of alcohol.
9. Patients receiving antiresorptive drugs such as bisphosphonates, denosumab, romosozumab or other drugs associated with osteonecrosis due to drugs such as m-TOR inhibitors, bevacizumab and sunitinib.
10. Pregnant or breastfeeding women.
11. Presence of oral lesions on the palate such as recurrent lesions due to herpes simplex virus.
12. Patients who use removable dental prosthesis that covers the palate.
13. Patients with a history of hypersensitivity to any of the materials used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction assessed by the Visual Analog Scale in the palate | day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 10, day 14
  Visual analog escale from 0 (the minimun and best score) to 10 (the maximum and worst pain score)
Satisfaction assessed by analgesic pills consumption | day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 10, day 14
  Number of Ibuprofens 600mg every 8hours (if needed) taken

SECONDARY OUTCOMES:
Satisfaction assessed by Oral Health Impact Profile 14 (OHIP-14) | day 0, day 3, day 7, day 14
  OHIP-14 questionnaire: 0 means the best score and 56 the maximum and worst score
Hematoma assessed by the patient | Assessed day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10 after the surgery
  yes / no
Swelling assessed by the patient | Assessed day 1, day 2, day 3,day 4, day 5, day 6, day 7, day 10,day 14 after the surgery
  yes / no
Palate bleeding assessed by the patient | Assessed before and after 24 hours postoperatively
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Rosa López-Pintor, Professor, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Clinica Dental Doctores Garcia Ruiz e Iglesias Esquiroz, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Moreno S, Lopez-Pintor RM, Leco-Berrocal I, Torres J, Gonzalez-Serrano J. Impact of a Bioadhesive Oral Wound Dressing Combined With Flowable Resin on Patient-Reported Outcomes After Palatal Graft Harvesting: A Randomized Clinical Trial. Clin Oral Implants Res. 2025 Nov 10. doi: 10.1111/clr.70070. Online ahead of print. PMID 41212657